CLINICAL TRIAL: NCT02075515
Title: Consistency, Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults 50 Years of Age or Older
Brief Title: Consistency, Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster (HZ) Vaccine GSK1437173A in Adults ≥ 50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 117177; 2013-000373-76 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: Safety; Zoster; Immunogenicity; Adults; Consistency
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- HZ/su Lot A (Experimental): Subjects will receive Lot A of the HZ/su vaccine at 0 and 2 months. The HZ/su vaccine composed of unique randomized combinations of an adjuvant lot and one gE lot.
  Interventions: Biological: Herpes Zoster vaccine (GSK 1437173A)
- HZ/su Lot B (Experimental): Subjects will receive Lot B of the HZ/su vaccine at 0 and 2 months. The HZ/su vaccine composed of unique randomized combinations of an adjuvant lot and one gE lot.
  Interventions: Biological: Herpes Zoster vaccine (GSK 1437173A)
- HZ/su Lot C (Experimental): Subjects will receive Lot C of the HZ/su vaccine at 0 and 2 months. The HZ/su vaccine composed of unique randomized combinations of an adjuvant lot and one gE lot.
  Interventions: Biological: Herpes Zoster vaccine (GSK 1437173A)

INTERVENTIONS:
Biological: Herpes Zoster vaccine (GSK 1437173A) — 2 doses administered intramuscularly in deltoid region of non-dominant arm.
  Other Names: HZ/su vaccine

SUMMARY:
The purpose of this study is to demonstrate lot-to-lot consistency in terms of immunogenicity, and evaluate safety of the Herpes Zoster subunit (HZ/su) vaccine. The study is designed as a randomized, double-blind study with three parallel groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female aged 50 years or older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. A prednisone dose of < 20 mg/day is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine (E.g. inactivated and subunit vaccines) within 8 days prior to or within 14 days after either dose of study vaccine.
* Administration of long-acting immune-modifying drugs within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against HZ or varicella.
* Planned administration during the study of an HZ or varicella vaccine other than the study vaccine.
* History of HZ.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C (99.5°F) on oral, axillary or tympanic route, or ≥ 38.0°C (100.4°F) on rectal route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating females.
* Females planning to become pregnant or planning to discontinue contraceptive precautions (if of childbearing potential) before Month 4.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Any condition which, in the judgment of the investigator would make intramuscular injection unsafe.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (3):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Milford, Massachusetts
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Wilrijk
- Canada (3):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Strezova A, Godeaux O, Aggarwal N, Leroux-Roels G, Lopez-Fauqued M, Van Damme P, Vanden Abeele C, Vastiau I, Heineman TC, Lal H. A randomized lot-to-lot immunogenicity consistency study of the candidate zoster vaccine HZ/su. Vaccine. 2017 Dec 4;35(48 Pt B):6700-6706. doi: 10.1016/j.vaccine.2017.10.017. Epub 2017 Oct 24. PMID 29079101
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1437173A Lot A Group: Male and female subjects, aged ≥ 50 years at the time of study vaccination, received a dose of the GSK1437173A vaccine from Lot A, administered intramuscularly in the deltoid region of non-dominant arm, at 0 and 2 months.
- GSK1437173A Lot B Group: Male and female subjects, aged ≥ 50 years at the time of study vaccination, received a dose of the GSK1437173A vaccine from Lot B, administered intramuscularly in deltoid region of non-dominant arm, at 0 and 2 months.
- GSK1437173A Lot C Group: Male and female subjects, aged ≥ 50 years at the time of study vaccination, received a dose of the GSK1437173A vaccine from Lot C, administered intramuscularly in deltoid region of non-dominant arm, at 0 and 2 months.
Period: Overall Study
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Started | 218 | 217 | 216
Completed | 214 | 212 | 208
Not Completed | 4 | 5 | 8
Not completed — Serious Adverse Event | 1 | 1 | 1
Not completed — Non-Serious Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- GSK1437173A Lot A Group: Male and female subjects, aged ≥ 50 years at the time of study vaccination, received a dose of the GSK1437173A vaccine from Lot A, administered intramuscularly in deltoid region of non-dominant arm, at 0 and 2 months.
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group | Total
Number analyzed (Participants) | 218 | 217 | 216 | 651
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (8.8) | 64.3 (9.4) | 64.4 (8.8) | 64.5 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 130 | 114 | 360
  Male | 102 | 87 | 102 | 291

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-gE Antibody Concentrations Equal to or Above the Cut-off Value
Description: Anti-gE antibody concentrations, as determined by Enzyme-linked Immunosorbent Assay (ELISA). The cut-off value was ≥ 97 milli international units per milliliter (mIU/mL).
Time Frame: At Month 3
Population: The analysis was performed on the according-to-protocol (ATP) cohort for immunogenicity, which included all eligible subjects who had post-vaccination immunogenicity results and who complied with the protocol, including the time schedule for vaccination and blood sample draw.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 210 | 210 | 202
Subjects | 210 | 210 | 202
Statistical Analysis 1: Comparison: GSK1437173A Lot A Group vs GSK1437173A Lot B Group; Test type: Non-Inferiority or Equivalence — Superiority Criterion: The two-sided 95 % CI of the GMC ratio between all pairs of lots are within [0.67, 1.5]; ANCOVA; Adjusted GMC Ratio = 0.97, 95% CI 2-sided [0.86 to 1.09]
Statistical Analysis 2: Comparison: GSK1437173A Lot A Group vs GSK1437173A Lot C Group; Test type: Non-Inferiority or Equivalence — Superiority Criterion: The two-sided 95 % CI of the GMC ratio between all pairs of lots are within [0.67, 1.5]; ANCOVA; Adjustd GMC Ratio = 0.96, 95% CI 2-sided [0.85 to 1.08]
Statistical Analysis 3: Comparison: GSK1437173A Lot B Group vs GSK1437173A Lot C Group; Test type: Non-Inferiority or Equivalence — Superiority Criterion: The two-sided 95 % CI of the GMC ratio between all pairs of lots are within [0.67, 1.5]; ANCOVA; Adjusted GMC ratio = 0.99, 95% CI 2-sided [0.88 to 1.10]

2. Secondary Outcome: Anti-gE Humoral Immunogenicity
Description: Anti-gE antibody concentrations, were determined by ELISA, expressed as Geometric Mean Concentrations (GMCs), in milli international units per milliliter (mIU/mL).
Time Frame: At Month 0 and Month 3
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all eligible subjects who had post-vaccination immunogenicity results and who complied with the protocol, including the time schedule for vaccination and blood sample draw.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 210 | 210 | 202
mIU/mL
  Anti-gE, Month 0 | 1378.4 [1180.0 to 1610.0] | 1166.5 [1005.5 to 1353.4] | 1381.2 [1190.9 to 1601.9]
  Anti-gE, Month 3 | 59556.1 [54587.6 to 64976.7] | 60733.8 [55995.2 to 65873.3] | 62058.3 [57422.3 to 67068.7]

3. Secondary Outcome: Number of Vaccine Responders for Anti-gE Concentrations as Determined by ELISA
Description: Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL); For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 210 | 210 | 202
Subjects | 201 | 205 | 197

4. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, that prevented normal every day activities.
Time Frame: Within 7 days (Days 0-6) after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered, only on those subjects with the symptoms sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 217 | 217 | 215
Subjects
  Any Pain, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Any Pain, Dose 1 | 160 | 179 | 166
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Grade 3 Pain, Dose 1 | 4 | 6 | 7
  Any Redness, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Any Redness, Dose 1 | 29 | 48 | 41
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Grade 3 Redness, Dose 1 | 1 | 1 | 1
  Any Swelling, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Any Swelling, Dose 1 | 24 | 33 | 26
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 217 | 217 | 214
  Grade 3 Swelling, Dose 1 | 0 | 0 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Any Pain, Dose 2 | 155 | 152 | 155
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Grade 3 Pain, Dose 2 | 18 | 13 | 7
  Any Redness, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Any Redness, Dose 2 | 38 | 47 | 43
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Grade 3 Redness, Dose 2 | 3 | 2 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Any Swelling, Dose 2 | 22 | 28 | 25
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 211 | 216 | 207
  Grade 3 Swelling, Dose 2 | 3 | 1 | 1
  Any Pain, Across Doses | 188 | 196 | 185
  Grade 3 Pain, Across Doses | 22 | 16 | 13
  Any Redness, Across Doses | 52 | 68 | 62
  Grade 3 Redness, Across Doses | 4 | 3 | 3
  Any Swelling, Across Doses | 38 | 44 | 39
  Grade 3 Swelling, Across Doses | 3 | 1 | 2

5. Secondary Outcome: Number of Days With Any Solicited Local Symptoms
Description: The number of days with any local symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7 days (Days 0-6) after each vaccine dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered and with results available for this assessment.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 217 | 217 | 215
Days
  Pain post-Dose 1 | 2.0 [2.0 to 3.5] | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 4.0]
  Pain post-Dose 2 | 2.0 [2.0 to 4.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Redness post-Dose 1 | 2.0 [2.0 to 3.0] | 3.0 [1.5 to 3.0] | 2.0 [2.0 to 4.0]
  Redness post-Dose 2 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
  Swelling post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 3.0 [2.0 to 4.0]
  Swelling post-Dose 2 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.0]

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal (nausea, vomiting, diarrhea and/or abdominal pain), headache, myalgia, shivering and temperature [defined as oral temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature= temperature > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 7 days (Days 0-6) after each vaccine dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered, only on those subjects with the symptom sheets filled in.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 217 | 217 | 216
Subjects
  Any Fatigue, Dose 1 | 66 | 68 | 64
  Grade 3 Fatigue, Dose 1 | 5 | 4 | 4
  Related Fatigue, Dose 1 | 62 | 63 | 58
  Any Gastrointestinal, Dose 1 | 23 | 22 | 26
  Grade 3 Gastrointestinal, Dose 1 | 1 | 0 | 4
  Related Gastrointestinal, Dose 1 | 19 | 20 | 23
  Any Headache, Dose 1 | 63 | 68 | 49
  Grade 3 Headache, Dose 1 | 5 | 4 | 4
  Related Headache, Dose 1 | 59 | 63 | 43
  Any Myalgia, Dose 1 | 85 | 89 | 76
  Grade 3 Myalgia, Dose 1 | 4 | 3 | 4
  Related Myalgia, Dose 1 | 71 | 78 | 62
  Any Shivering, Dose 1 | 31 | 21 | 22
  Grade 3 Shivering, Dose 1 | 1 | 4 | 0
  Related Shivering, Dose 1 | 30 | 19 | 21
  Any Temperature, Dose 1 | 28 | 23 | 22
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0
  Related Temperature, Dose 1 | 24 | 21 | 19
  Any Fatigue, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Fatigue, Dose 2 | 91 | 85 | 82
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Fatigue, Dose 2 | 14 | 7 | 6
  Related Fatigue, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Fatigue, Dose 2 | 89 | 80 | 76
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Gastrointestinal, Dose 2 | 33 | 34 | 29
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Gastrointestinal, Dose 2 | 2 | 2 | 5
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Gastrointestinal, Dose 2 | 29 | 29 | 28
  Any Headache, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Headache, Dose 2 | 74 | 80 | 66
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Headache, Dose 2 | 9 | 11 | 5
  Related Headache, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Headache, Dose 2 | 69 | 76 | 63
  Any Myalgia, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Myalgia, Dose 2 | 99 | 91 | 83
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Myalgia, Dose 2 | 20 | 11 | 7
  Related Myalgia, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Myalgia, Dose 2 | 85 | 81 | 76
  Any Shivering, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Shivering, Dose 2 | 67 | 60 | 44
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Shivering, Dose 2 | 11 | 5 | 7
  Related Shivering, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Shivering, Dose 2 | 66 | 59 | 43
  Any Temperature, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Any Temperature, Dose 2 | 43 | 34 | 25
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Grade 3 Temperature, Dose 2 | 2 | 0 | 1
  Related Temperature, Dose 2: number analyzed (Participants) | 212 | 216 | 208
  Related Temperature, Dose 2 | 40 | 33 | 25
  Any Fatigue, Across Doses | 114 | 109 | 107
  Grade 3 Fatigue, Across Doses | 18 | 11 | 10
  Related Fatigue, Across Doses | 111 | 102 | 103
  Any Gastrointestinal, Across Doses | 46 | 45 | 50
  Grade3 Gastrointestinal,Across Doses | 3 | 2 | 9
  Any Headache, Across Doses | 101 | 108 | 89
  Grade 3 Headache, Across Doses | 13 | 13 | 9
  Related Headache, Across Doses | 95 | 101 | 82
  Any Myalgia, Across Doses | 128 | 119 | 113
  Grade 3 Myalgia, Across Doses | 24 | 12 | 10
  Related Myalgia, Across Doses | 112 | 107 | 102
  Any Shivering, Across Doses | 80 | 67 | 60
  Grade 3 Shivering, Across Doses | 12 | 7 | 7
  Related Shivering, Across Doses | 79 | 65 | 58
  Any Temperature, Across Doses | 59 | 49 | 43
  Grade 3 Temperature, Across Doses | 2 | 0 | 1
  Related Temperature, Across Doses | 53 | 46 | 41
  Related Gastrointestinal, Across Doses | 41 | 39 | 46

7. Secondary Outcome: Number of Days With Any Solicited General Symptoms
Description: The number of days with any general symptoms reported during the solicited post-vaccination period.
Time Frame: During the 7 days (Days 0-6) after each vaccine dose
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 217 | 217 | 216
Days
  Fatigue post-Dose 1 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue post-Dose 2 | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Gastrointestinal symptoms post-Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Gastrointestinal symptoms post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Headache post-Dose 1 | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Myalgia post-Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Myalgia post-Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Shivering post-Dose 1 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering post-Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 2.0]
  Temperature post-Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Temperature post-Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]

8. Secondary Outcome: Number of Subjects With Any Potential Immune-Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology
Time Frame: From first vaccination up to 30 days post last vaccination (Month 0-Month 3) and from Month 4 until study end (Month 14)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one dose of the study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 218 | 217 | 216
Subjects
  pIMDs from Month 0 to Month 3 | 3 | 0 | 1
  pIMDs from Month 4 to Month 14 | 2 | 0 | 2

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During 30 days (Days 0-29) after each vaccination
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 218 | 217 | 216
Subjects
  Any AE(s) | 72 | 69 | 76
  Grade 3 AE(s) | 13 | 15 | 9
  Related AE(s) | 23 | 22 | 27

10. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From first vaccination up to 30 days post last vaccination (Month 0-Month 3) and from Month 4 to study end (Month 14)
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Number analyzed (Participants) | 218 | 217 | 216
Subjects
  SAEs from Month 0 to Month 3 | 5 | 7 | 4
  SAEs from Month 4 to Month 14 | 10 | 8 | 16

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: within 7 days (Days 0-6) after each vaccination; Unsolicited AEs: during 30 days (Days 0-29) after each vaccination; SAEs: from first vaccination up to study end (Month 0-Month 14).
Arm/Group | GSK1437173A Lot A Group | GSK1437173A Lot B Group | GSK1437173A Lot C Group
Serious Adverse Events (participants affected / at risk) | 13/218 | 14/217 | 20/216
Other Adverse Events (participants affected / at risk) | 202/218 | 201/217 | 198/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1437173A Lot A Group (N=218) | GSK1437173A Lot B Group (N=217) | GSK1437173A Lot C Group (N=216)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 0 | 1 | 0
Pancreas infection (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1437173A Lot A Group (N=218) | GSK1437173A Lot B Group (N=217) | GSK1437173A Lot C Group (N=216)
Gastrointestinal disorder (Gastrointestinal disorders) | 46 | 45 | 50
Chills (General disorders) | 80 | 67 | 61
Fatigue (General disorders) | 114 | 109 | 107
Pain (General disorders) | 188 | 196 | 185
Pyrexia (General disorders) | 60 | 50 | 43
Swelling (General disorders) | 38 | 44 | 40
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 128 | 119 | 113
Headache (Nervous system disorders) | 101 | 108 | 89
Erythema (Skin and subcutaneous tissue disorders) | 55 | 70 | 62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.